CLINICAL TRIAL: NCT02481739
Title: Study of the Impact of Laparoscopic Surgical Management of Endometriosis on Fertility
Brief Title: Laparoscopic Surgical Management of Endometriosis on Fertility
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6201
Record Dates: First submitted 2015-06-07; First posted 2015-06-25 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2015-06

CONDITIONS: Endometriosis
Keywords: endometriosis; fertility; endometriosis surgery
MeSH Terms: conditions — Endometriosis | interventions — Retrospective Studies

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: retrospective study

SUMMARY:
The aim of the investigators study is to know the results of the endometriosis surgery and particularly to highlight a benefit of this surgery on fertility.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Patients operated by laparoscopy for endometriosis in our department between 2006 and 2014.

Exclusion Criteria:

* Patients under 18 years

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This work concerns patients aged 18-38 years, operated by laparoscopy for endometriosis in our department between 2006 and 2014
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
benefit of endometriosis surgery on fertility : occurrence of pregnancy or live birth, spontaneous or after use of a MPA technical | after surgery, up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud WATTIEZ, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Service de Gynécologie, Strasbourg, France, France